CLINICAL TRIAL: NCT02951650
Title: Long Term Observational Study of the Safety and Efficacy of an Active Implantable Vagal Nerve Stimulation Device in Patients With Crohn's Disease
Brief Title: Long Term Observational Study of a Vagal Nerve Stimulation Device in Crohn's Disease
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: SetPoint Medical Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPM-010
Record Dates: First submitted 2016-10-29; First posted 2016-11-01 (Estimated); Last update posted 2017-08-03 (Actual); Status verified 2017-08

CONDITIONS: Crohn Disease
Keywords: vagus nerve stimulation
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cyberonics VNS (Experimental): Cyberonics VNS
  Interventions: Device: Cyberonics VNS

INTERVENTIONS:
Device: Cyberonics VNS — Vagus nerve stimulation

SUMMARY:
This will be an open label multicenter study of the safety and efficacy of an active implantable VNS device in patients with Crohn's Disease.

DETAILED DESCRIPTION:
Patients who complete study SPM-007 will be enrolled in this study at the time of the last visit of the preceding study. The assessments at the last visit of the preceding study will also be used as baseline measures for the current study. If the patient has previously discontinued SPM-007 and greater than 30 days have elapsed since the final visit in SPM-007, baseline measures for the current study will be repeated, and an interim medical history will be taken to assess whether any new medical conditions were diagnosed in the time between studies.

The study will continue until the last patient entered has completed 24 months in this study.

Follow-up visits will occur at 3, 6, 12, 18 and 24 months. A final follow-up visit will occur for all remaining patients at study closure when the final enrolled subject has completed 24 months on study.

An Interim Visit must be performed a maximum of 1 month after any change in device settings. Interim visits may also be performed at any time at the principal investigator's discretion; either between scheduled visits, or after the patient has completed the Month 24 Visit, if the study is still ongoing.

ELIGIBILITY:
Inclusion Criteria:

Patients must have enrolled in study SPM-007; including patients who either completed that study or withdrew before completion of that study.

Exclusion Criteria:

Inability to provide informed consent Significant psychiatric illness or substance abuse

All patients will be excluded who have developed any of these exclusionary conditions during the SMP-007 study, or in the interim between SPM-007 and the Day 0 of SPM-010:

* History of unilateral or bilateral vagotomy
* History of recurrent vaso-vagal syncope episodes
* Known obstructive sleep apnea
* Known history of cardiac rhythm disturbances, atrio-ventricular block of greater than first degree, or cardiac conduction pathway abnormalities other than isolated right bundle branch block or isolated left anterior fascicle block.
* Significant pharyngeal dysfunction or swallowing difficulties
* Clinically significant vocal cord damage or hoarseness
* Other implanted electrically active medical devices (e.g., cardiac pacemakers, automatic implantable cardioverter-defibrillators)
* Asthma or chronic obstructive pulmonary disease not controlled by medications, or any other disease causing clinically significant dyspnea
* A greater than or equal to 40 pack-year smoking history
* Active peptic ulcer disease
* Patients with a limited life expectancy due to terminal illness

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2015-01; Primary Completion 2018-05 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
Crohn's Disease Activity Index | 24 months

SECONDARY OUTCOMES:
Inflammatory Bowel Disease Questionnaire | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Geert D'Haens, M.D., Ph.D., Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (4):
- Dubrava Hospital, Zagreb, Croatia
- Humanitas Research Hospital, Milan, Italy
- Academic Medical Center, Amsterdam, Netherlands
- Karolinska Institute, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No